CLINICAL TRIAL: NCT01183234
Title: Phase 1,Randomized,Open-Label,Two Period Single Dose Crossover Bioequivalence Study of Two Capsule Strengths of SPD544 In Healthy Volunteers.
Brief Title: SPD544 High Strength Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPD544-101
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Results first posted 2011-08-25 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPD544 (Equasym XL) (Experimental)
  Interventions: Drug: SPD544
- Methylphenidate hydrochloride (Metadate CD ) (Experimental)
  Interventions: Drug: Methylphenidate hydrochloride

INTERVENTIONS:
Drug: SPD544 — two 30mg capsules, single oral dose
  Other Names: Equasym XL
  Arms: SPD544 (Equasym XL)
Drug: Methylphenidate hydrochloride — one 60mg capsule, single oral dose
  Other Names: Metadate CD
  Arms: Methylphenidate hydrochloride (Metadate CD )

SUMMARY:
The purpose of this study is to assess bioequivalence of 2 capsule strengths.

DETAILED DESCRIPTION:
This will be a randomised, open-label, two-period, single dose, crossover bioequivalence study in healthy subjects under fasting conditions to assess bioequivalence of 1 x 60 mg capsule methylphenidate compared to 2 x 30 mg capsules methylphenidate. Pharmacokinetics and safety will be assessed.

ELIGIBILITY:
Inclusion criteria:

1. Healthy subjects, aged 18-55 years inclusive at the time of consent.
2. Subject must be willing to comply with applicable contraceptive requirements of the protocol and be:

   * Male, or
   * Non-pregnant, non-lactating female who must be >90 days post-partum or nulliparous.
3. Body Mass Index (BMI) between 18.5 and 30.0kg/m² inclusive. This inclusion criterion will only be assessed at the Screening visit.
4. Satisfactory medical assessment with no clinically significant or relevant abnormalities in medical history, physical examination, vital signs, ECG, and clinical laboratory evaluation (haematology, biochemistry, urinalysis) as assessed by the Investigator.
5. Ability to provide written, personally signed and dated informed consent to participate in the study.
6. An understanding, ability and willingness to fully comply with study procedures and restrictions.
7. Ability to swallow all investigational medicinal products (IMPs).

Exclusion criteria:

1. Current or recurrent disease (e.g., cardiovascular, renal, liver, gastrointestinal, malignancy or other conditions) that could affect the action, absorption, or disposition of the IMPs, or could affect clinical or laboratory assessments.
2. Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the IMPs or study procedures.
3. Current use of any medication (including prescription, over-the-counter [OTC], herbal, or homeopathic preparations) with the exception of hormone replacement therapy or hormonal contraceptives and/or an occasional dose of nonsteroidal anti-inflammatory (NSAID), or paracetamol (current use is defined as use within 14 days of first dose of IMP).
4. History of hypertension or a resting sitting systolic blood pressure >139mmHg or diastolic blood pressure >89mmHg.
5. History of seizure (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or family history of Tourette's Disorder.
6. Known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, transient ischaemic attack or stroke, or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
7. Family history of sudden cardiac death or ventricular arrhythmia.
8. Known cerebrovascular disorders such as cerebral aneurysm, vascular abnormalities including vasculitis or history of stroke.
9. Diagnosis of glaucoma.
10. Diagnosis of phaeochromocytoma.
11. Current abnormal thyroid function, as defined as abnormal screening thyroid stimulating hormone (TSH) and thyroxine (T4).
12. Current marked anxiety, tension and/or agitation.
13. History of alcohol or other substance abuse within the last year.
14. A positive screen for alcohol or drugs of abuse at Screening or Day -1 of Treatment Period 1.
15. Male subjects who consume more than 3 units of alcohol per day. Female subjects who consume more than 2 units of alcohol per day.
16. A positive human immunodeficiency virus (HIV) antibody screen, Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibody screen.
17. Use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch) within 30 days prior to the Screening visit.
18. Routine consumption of more than 300mg of caffeine per day or subjects who experience caffeine withdrawal headaches or have a history of caffeine withdrawal headaches.
19. Donation of blood or blood products (e.g., plasma or platelets) within 90 days prior to the first dose of IMP.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-08-27 (Actual); Primary Completion 2010-10-22 (Actual); Study Completion 2010-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Paraxel International, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Equasym XL (SPD544) First, Then Metadate CD: Subjects received a single oral dose of 60 mg of Equasym XL (given as two 30 mg capsules), then a 7-day washout period, then subjects received a single oral dose of 60 mg of Metadate CD (given as one 60 mg capsule)
- Metadate CD First, Then Equasym XL: Subjects received a single oral dose of 60 mg of Metadate CD (given as one 60 mg capsule), then a 7-day washout period, then subjects received a single oral dose of 60 mg of Equasym XL (given as two 30 mg capsules)
Period: First Intervention
Arm/Group | Equasym XL (SPD544) First, Then Metadate CD | Metadate CD First, Then Equasym XL
Started | 14 | 14
Completed | 13 | 14
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout
Arm/Group | Equasym XL (SPD544) First, Then Metadate CD | Metadate CD First, Then Equasym XL
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Equasym XL (SPD544) First, Then Metadate CD | Metadate CD First, Then Equasym XL
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Equasym XL First, Then Metadate CD: Subjects received a single oral dose of 60 mg of Equasym XL (SPD544, Methylphenidate HCl given as two 30 mg capsules), then a 7-day washout period, then subjects received a single oral dose of 60 mg of Metadate CD (Methylphenidate HCl given as one 60 mg capsule)
- Metadate CD First, Then Equasym XL: Subjects received a single oral dose of 60 mg of Metadate CD (Methylphenidate HCl given as one 60 mg capsule), then a 7-day washout period, then subjects received a single oral dose of 60 mg of Equasym XL (SPD544, Methylphenidate HCl given as two 30 mg capsules)
- Total: Total of all reporting groups
Arm/Group | Equasym XL First, Then Metadate CD | Metadate CD First, Then Equasym XL | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Customized [Mean (Standard Deviation); unit: years] | 30.8 (10.12) | 29.5 (8.61) | 30.1 (9.24)
Age, Customized [Count of Participants; unit: Participants]
  18 to 55 years | 14 | 14 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 10 | 7 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC 0-t) for Methylphenidate Hydrochloride (MPH) Using Two Different Formulations (Equasym XL and Metadate CD)
Description: AUC 0-t is the area under the plasma concentration versus time curve from time 0 to the time of last quantifiable concentration. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: predose and 0.5, 1.0, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20 and 24 hours post-dose
Population: Pharmacokinetic analysis set (PK) defined as all subjects in the safety analysis set who had evaluable plasma concentration-time profiles for MPH through 24 hours post-dosing in both treatment periods. Subjects who vomited or experienced significant diarrhea between dosing and 10 hours post-dose were excluded.
Measure: Least Squares Mean (90% Confidence Interval); unit: ng*h/ml
Groups:
- Equasym XL: Subjects received a single oral dose of 60 mg of Equasym XL (Methylphenidate HCl given as two 30 mg capsules)
- Metadate CD: Subjects received a single oral dose of 60 mg of Metadate CD (Methylphenidate HCl given as one 60 mg capsule)
Arm/Group | Equasym XL | Metadate CD
Number analyzed (Participants) | 27 | 27
ng*h/ml | 133 [122 to 145] | 127 [116 to 138]
Statistical Analysis 1: Comparison: Equasym XL vs Metadate CD; Test type: Non-Inferiority or Equivalence — Point estimates and 90% confidence intervals for the ratio of the treatment regimen means were provided by back-transformation on to the linear scale and were assessed against the currently accepted bioequivalence criteria for log-transformed data (0.80, 1.25); Mixed Models Analysis; Ratio of geometric LS means = 0.953, 90% CI 2-sided [0.915 to 0.993]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) for MPH Using Two Different Formulations (Equasym XL and Metadate CD)
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: predose and 0.5, 1.0, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20 and 24 hours post-dose
Population: PK set
Measure: Least Squares Mean (90% Confidence Interval); unit: ng/ml
Arm/Group | Equasym XL | Metadate CD
Number analyzed (Participants) | 27 | 27
ng/ml | 14.9 [13.8 to 16.1] | 14.7 [13.7 to 15.9]
Statistical Analysis 1: Comparison: Equasym XL vs Metadate CD; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of geometric LS means = 0.988, 90% CI 2-sided [0.931 to 1.05]

3. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) for MPH Using Two Different Formulations (Equasym XL and Metadate CD)
Description: Tmax is the time after administration of a drug when the maximum plasma concentration in the body is reached.
Time Frame: predose and 0.5, 1.0, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20 and 24 hours post-dose
Population: PK set
Measure: Median (Full Range); unit: hours
Arm/Group | Equasym XL | Metadate CD
Number analyzed (Participants) | 27 | 27
hours | 5.0 [0.983 to 5.15] | 5.0 [0.967 to 6.05]
Statistical Analysis 1: Comparison: Equasym XL vs Metadate CD; Test type: Superiority or Other; Wilcoxon (Hodges-Lehmann); Median Difference (Final Values) = 0.0, 90% CI 2-sided [-0.150 to 0.492]

ADVERSE EVENTS:
Description: Safety Analysis Set consisted of subjects who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Arm/Group | Equasym XL | Metadate CD
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 10/28 | 6/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Equasym XL (N=28) | Metadate CD (N=27)
Dry mouth (Gastrointestinal disorders) | 5 | 3
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually